CLINICAL TRIAL: NCT04213989
Title: An Investigator-initiated Study Assessing the Effect of Intermittent Pneumatic Compression (IPC) on Symptoms and Quality of Life in Women With Lipo-lymphedema (Lipedema With Swelling)
Brief Title: Intermittent Pneumatic Compression in Women With Lipo-lymphedema (Lipedema With Swelling)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Wright, MD (Industry)
Collaborators: Tactile Medical (Industry)
Responsible Party: Sponsor-Investigator, Thomas Wright, MD, MD, FACPh, FACP, RVT, Tactile Medical
Organization: Tactile Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000
Record Dates: First submitted 2019-12-21; First posted 2019-12-30 (Actual); Results first posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Lipedema; Lipolymphedema
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to conservative care or Flexitouch Plus and conservative care at Screening. Subjects have up to 60 days to acquire treatment through commercial means and commence treatment. Follow-up will take place 3-4 weeks after treatment commences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conservative Care (Active Comparator): Conservative care (may include 30-40 mmHg graduated compression up to waist, dietary counseling, exercise, and/or referral for CDT)
  Interventions: Other: Conservative Care
- Flexitouch Plus and Conservative Care (Experimental): Flexitouch Plus with conservative care
  Interventions: Device: Flexitouch Plus and Conservative Care

INTERVENTIONS:
Device: Flexitouch Plus and Conservative Care — A segmental, programmable, gradient advanced pneumatic compression device. The system consists of a controller unit and garments, and provides in-home manual lymphatic drainage therapy in the legs for approximately 1 hour daily. Conservative care may include 30-40 mmHg graduated compression up to waist, dietary counseling, exercise, and/or referral for CDT.
  Other Names: Flexitouch system
  Arms: Flexitouch Plus and Conservative Care
Other: Conservative Care — May include 30-40 mmHg graduated compression up to waist, dietary counseling, exercise, and/or referral for CDT.
  Arms: Conservative Care

SUMMARY:
Lipedema is a connective tissue disorder that affects up to 10% of women. It is characterized by painful, swollen subcutaneous tissue and disproportionate fat accumulation (primarily in the lower limbs, however it can spread to the abdomen and arms). Patients are often not aware they are affected by this disease; rather, they think they are just overweight or obese.

Patients with lipedema often feel frustrated and uncomfortable as symptoms such as heaviness, pain, and easy bruising impact quality of life. Affected limbs can become so large and heavy that daily tasks such as walking, cleaning, or shopping become impossible.

There is currently no cure for lipedema, thus treatment focuses on symptom management and improved patient-reported outcomes. At present, the two main courses of treatment include non-surgical conservative treatment (e.g., Comprehensive Decongestive Therapy (CDT), diet, exercise, emotional/psychological/social support) and lymph-sparing liposuction performed by a surgeon trained in lipedema treatment. The primary goals for treatment include: reduction/elimination of inflammation, swelling, and pain; increase in lymphatic flow, which reduces/eliminates excessive fluid and swelling; overall management of the physical impact of lipedema; and quality of life improvements which can include emotional, psychological/mental, spiritual, and social enhancement in addition to physical management.

Intermittent Pneumatic Compression (IPC) devices are often used as home-therapy to treat secondary lymphedema or lipo-lymphedema (lipedema with swelling) and may be helpful in preventing the progression of lipedema. IPC use moves lymphatic fluid and supports the elimination of proteinaceous fluids, thus leading to improved patient-reported symptoms, decreased limb girth and volume, increased elasticity of tissues, and fewer episodes of infection.

The purpose of this study is to assess whether 3-4 weeks of IPC usage is associated with alleviation of symptoms and improvement in quality of life in women with lipo-lymphedema (lipedema with swelling).

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-70 years
* Stage 2-3 (Schmeller Type 2-3) lipedema with secondary lymphedema
* Willing and able to follow prescribed care for study period
* Able to access (via self-pay, patient assistance, or insurance programs) prescribed care within 60 days of Screening visit

Exclusion Criteria:

* BMI > 50
* Heart failure (acute pulmonary edema, decompensated acute heart failure)
* Pacemaker or implantable cardioverter defibrillator (ICD)
* Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)
* Severe peripheral artery disease (critical limb ischemia including ischemic rest pain, arterial wounds, or gangrene)
* Active skin or limb infection/inflammatory disease (acute cellulitis, other uncontrolled skin or untreated inflammatory skin disease) on the arms or trunk
* Active cancer (cancer that is currently under treatment, but not yet in remission)
* Poorly controlled kidney disease (glomerular filtration rate < 30 mls per minute), hypoproteinemia, pulmonary hypertension, hypothyroidism, cyclic edema, or Munchausen Syndrome
* Any circumstance where increased lymphatic or venous return is undesirable
* Currently pregnant or trying to become pregnant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wright, MD, Principal Investigator — Lakeview Medical Group, Inc
Locations (1):
- Laser Lipo and Vein Center, O'Fallon, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Started | 18 | 18
Completed | 14 | 12
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (9.6) | 44.6 (9.5) | 43.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26
BMI [Mean (Standard Deviation); unit: kg/m^2] | 37.0 (7.5) | 35.9 (5.2) | 36.5 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Circumferential Measurements Over Time
Description: Tape measurements along both legs
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Measure: Mean (95% Confidence Interval); unit: cm
Units Other Than Participants: Legs
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
Number analyzed (Legs) | 28 | 24
cm
  Ankle | -0.5 [-0.9 to -0.1] | -1.0 [-1.4 to -0.5]
  Calf | -1.3 [-1.9 to -0.6] | -2.0 [-2.7 to -1.2]
  Knee | -2.4 [-3.7 to -1.2] | -4.7 [-6.0 to -3.4]
  Thigh | -1.7 [-2.7 to -0.8] | -3.0 [-4.1 to -2.0]
  Hip | -0.4 [-4.7 to 3.9] | 3.2 [-1.5 to 7.9]
  Waist | -2.4 [-4.0 to -0.7] | -2.3 [-4.1 to -0.5]

2. Primary Outcome: Patient-Reported Quality of Life
Description: RAND 36-Item Short Form Survey Instrument (SF-36) 1.0 is a global assessment of health impacts on quality of life that taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
score on a scale
  General health | -2.7 [-10.9 to 5.5] | 1.3 [-7.6 to 10.2]
  Physical functioning | 2.6 [-3.7 to 8.9] | 5.3 [-1.5 to 12.1]
  Role limitations due to physical functioning | -1.2 [-21.9 to 19.5] | 1.4 [-20.9 to 23.8]
  Emotional wellbeing | 2.8 [-1.9 to 7.6] | -1.0 [-6.1 to 4.2]
  Role limitations due to emotional problems | -10.9 [-26.7 to 4.8] | -2.2 [-18.5 to 14.3]
  Energy/fatigue | 4.8 [-2.2 to 11.8] | 0.7 [-6.9 to 8.3]
  Social functioning | 9.9 [-0.2 to 20.0] | -2.2 [-13.1 to 8.7]
  Pain | 4.5 [-2.1 to 11.0] | 10.2 [3.1 to 17.3]

3. Primary Outcome: Patient-Reported Pain Interference
Description: PROMIS Item Bank v1.0 - Pain Interference - Short Form 6b is a 6 item survey that measures self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. All items are scored so that a low score is associated with less pain interference (a more favorable health state). In addition, each item is scored on a 1 to 5 range so that the lowest and highest possible scores are 6 and 30, respectively.
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
score on a scale | -1.4 [-4.8 to 2.1] | -3.0 [-6.8 to 0.7]

4. Primary Outcome: Patient-Reported Pain
Description: Wong Baker Faces Scale is a self-assessment tool that is easily understood by patients, so they are able to choose the face that best illustrates the physical pain they are experiencing associated with their lipo-lymphedema. Face 0 doesn't hurt at all. Face 2 hurts just a little bit. Face 4 hurts a little bit more. Face 6 hurts even more. Face 8 hurts a whole lot. Face 10 hurts as much as you can imagine, although you don't have to be crying to have this worst pain.
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
score on a scale | -0.8 [-1.7 to 0.0] | -0.8 [-1.8 to 0.1]

5. Primary Outcome: Patient-Reported Symptoms of Lipo-Lymphedema
Description: NRS Symptom Survey is a 6-item survey that asks patients to rate their perceptions of swelling, heaviness, pain, fatigue, tenderness, and tightness independently for each leg using a 10-point numerical rating scale where 0 represents none/not present and 10 is worst imaginable. All items are scored so that a low score is associated with fewer symptoms (defines a more favorable health state). The lowest and highest possible scores per leg are 0 and 60, respectively, with a combined total score between 0 and 120.
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
score on a scale
  Swelling-Left Leg | -0.5 [-1.7 to 0.8] | -0.2 [-1.6 to 1.2]
  Heaviness-Left Leg | -0.9 [-2.0 to 0.3] | -1.0 [-2.2 to 0.3]
  Pain-Left Leg | -0.3 [-1.4 to 0.9] | -1.4 [-2.6 to -0.1]
  Fatigue-Left Leg | -1.4 [-2.5 to -0.4] | -0.6 [-1.7 to 0.5]
  Tenderness-Left Leg | -0.6 [-1.7 to 0.6] | -0.2 [-1.4 to 1.0]
  Tightness-Left Leg | -1.2 [-2.1 to -0.2] | -1.8 [-2.9 to -0.8]
  Swelling-Right Leg | -0.7 [-1.8 to 0.4] | 0.1 [-1.2 to 1.3]
  Heaviness-Right Leg | -0.8 [-1.7 to 0.1] | -0.5 [-1.5 to 0.4]
  Pain-Right Leg | -0.1 [-1.2 to 1.1] | -0.5 [-1.8 to 0.8]
  Fatigue-Right Leg | -1.8 [-2.9 to -0.7] | -0.3 [-0.5 to 0.8]
  Tenderness-Right Leg | -0.1 [-1.2 to 1.0] | 0.1 [-1.1 to 1.3]
  Tightness-Right Leg | -0.9 [-2.0 to 0.2] | -1.6 [-2.7 to -0.4]

6. Secondary Outcome: Patient-Reported Mobility
Description: PROMIS Item Bank v2.0 - Mobility is a 15-item survey that focuses on activities of physical mobility such as getting out of bed or a chair to activities such as running. All items are scored so that a high score is associated with more mobility (a more favorable health state). In addition, each item is scored on a 5 to 1 range so that the highest and lowest possible scores are 75 and 15, respectively.
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
score on a scale | 2.9 [0.4 to 5.4] | -0.6 [-3.4 to 2.1]

7. Secondary Outcome: Change in Bioimpedance Measurements Over Time
Description: InBody 770 whole body and segmental extracorporeal body weight / total body weight ratios
Time Frame: Changes between Screening and 3-4 weeks will be assessed
Population: Each participant underwent circumferential measurement at baseline and at follow-up. Patients were measured at 4 sites on each leg (narrowest part of the ankle, largest part of the calf, top of knee cap, and thickest part of the upper thigh), the widest part of the hips and the widest part of the waist.
Measure: Mean (95% Confidence Interval); unit: ohms
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
Number analyzed (Participants) | 14 | 12
ohms
  Whole body | -0.001 [-0.004 to 0.001] | -0.002 [-0.005 to 0.000]
  Trunk | -0.001 [-0.003 to 0.001] | -0.002 [-0.005 to 0.000]
  Arms | 0.000 [-0.001 to 0.001] | 0.000 [-0.001 to 0.001]
  Legs | -0.003 [-0.005 to -0.000] | -0.004 [-0.006 to -0.002]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: This study collected data on serious and device-related adverse events only. Non-serious adverse events were not required to reported and / or moniotred.
Arm/Group | Conservative Care | Flexitouch Plus and Conservative Care
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04213989/Prot_SAP_000.pdf